CLINICAL TRIAL: NCT06685809
Title: A Phase 1 Study Assessing Safety, Tolerability, Pharmacokinetics and Physiological Response (Pain Tolerance) to Single and Multiple Ascending Doses of FZ008-145 in Healthy Subjects.
Brief Title: A Phase 1 Study of FZ008-145 in Healthy Subjects.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Fermion Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: FZ008-P101; CTR20240574 (Registry Identifier: JKN23061)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- FZ008-145 solution- Part A (Experimental): All participants will receive single dose of oral FZ008-145 solution or placebo.
  Interventions: Drug: FZ008-145 solution; Drug: Placebo
- FZ008-145 tablet- Part B (Experimental): All participants will receive single dose of oral FZ008-145 tablet or placebo.
  Interventions: Drug: FZ008-145 Tablet; Drug: Placebo
- FZ008-145 tablet - Part D (Experimental): Subjects will participate in a 3-period, 3-treatment, 6-sequence crossover study. Each subject will receive a single oral dose of FZ008-145 tablet at two different dose levels and placebo, with each treatment administered in a randomized sequence.
  Each treatment period will be separated by a washout period of at least 10 days. Cold pressor testing will be conducted following each dosing to assess pain tolerance.
  Interventions: Drug: FZ008-145 Tablet; Drug: Placebo
- FZ008-145 tablet - Part D2 (Experimental): Subjects will participate in a 3-period, 3-treatment, 6-sequence crossover study. Each subject will receive a higher single oral dose of FZ008-145 tablet at two h and placebo, with each treatment administered in a randomized sequence.
  Each treatment period will be separated by a washout period of at least 10 days. Cold pressor testing will be conducted following each dosing to assess pain tolerance.
  Interventions: Drug: FZ008-145 Tablet; Drug: Placebo
- FZ008-145 tablet - Part E (Experimental): Part E includes up to 6 cohorts (E1-E6). Subjects will be enrolled into 6 sequential cohorts. Each cohort will receive once-daily or twice daily oral doses of FZ008-145 or placebo tablet for 14 consecutive days under fasted conditions.
  Interventions: Drug: FZ008-145 Tablet; Drug: Placebo

INTERVENTIONS:
Drug: FZ008-145 solution — Dose formulation- Oral solution
  Other Names: FZ008-145 Oral solution
  Arms: FZ008-145 solution- Part A
Drug: FZ008-145 Tablet — Dose formulation- Oral tablet
  Other Names: FZ008-145 Oral tablet
  Arms: FZ008-145 tablet - Part D; FZ008-145 tablet - Part D2; FZ008-145 tablet - Part E; FZ008-145 tablet- Part B
Drug: Placebo — Dose formulation- Matching doses
  Other Names: Matching doses/form placebo

SUMMARY:
The study will be conducted in 5 parts: Part A (single ascending dose [SAD] in solution formulation), Part C (food effect [FE]), Part D (cold pressor test [CPT] to evaluate pain tolerance following single dose), and Part E (multiple ascending dose [MAD] in tablet formulation).

DETAILED DESCRIPTION:
* Part A is a randomized, double-blind, placebo-controlled, SAD study to assess safety, tolerability, and pharmacokinetics (PK) of FZ008-145 solution in healthy subjects. Up to 40 subjects will be enrolled in 5 cohorts.
* Part B is a randomized, double-blind, placebo-controlled, SAD study to assess safety, tolerability, and PK of FZ008-145 tablet in healthy subjects. Up to 72 subjects will be enrolled in 9 cohorts.
* Part D is a randomized, double-blind, placebo-controlled, 3-period, 3-treatment, 6-sequence crossover study to evaluate the cold pain tolerance effect of FZ008-145 tablet in healthy subjects. A total of 12 healthy subjects will be randomized to receive each of the three treatments (FZ008-145 at two dose levels and placebo) across three treatment periods, with appropriate washout between periods.
* Part D2 is a randomized, double-blind, placebo-controlled, 3-period, 3-treatment, 6-sequence crossover study to evaluate the cold pain tolerance effect of FZ008-145 tablet in healthy subjects. A total of 12 healthy subjects will be randomized to evaluates higher single oral doses (FZ008-145 at two dose levels and placebo) across three treatment periods, with appropriate washout between periods.
* Part E is an open-label, multiple ascending dose (MAD) study to assess the safety, tolerability, and pharmacokinetics of FZ008-145 tablet in healthy subjects. Approximately 48 healthy subjects will be enrolled into 6 sequential cohorts receiving once-daily or twice daily oral doses of FZ008-145 for 14 consecutive days under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
2. Male or female aged 18 to 65 years (inclusive).
3. Subject has body mass index of 18 to 32 kg/m2 with a minimum body weight of 50 kg for males, and 45 kg for females (inclusive).
4. Subject is generally healthy, in the opinion of the Investigator, based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and other relevant tests conducted at Screening, Day 1 for Part D/Part D2 (period 1) and Day -1 for other parts at the discretion of the Investigator or designee. Tests could be repeated once if they are outside the relevant clinical reference range.
5. Subject has clinical laboratory values (based on hematology, coagulation, biochemistry, and urinalysis parameters) within normal range, as specified by the testing laboratory, at Screening and Day -1 (for all parts except Part D/Part D2), unless deemed not clinically significant by the Investigator or delegate. Tests could be repeated once if they are outside the relevant clinical reference range.
6. Females must not be pregnant or lactating, and must use acceptable, highly effective double contraception from Screening until 90 days after study completion, including the Follow-up period. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day -1 and be willing to have additional pregnancy tests as required throughout the study. Women not of childbearing potential must be postmenopausal for ≥ 12 months (postmenopausal status is to be confirmed through testing of follicle stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female subjects). Females must not donate eggs from the first dose of IP until at least 90 days after the last dose of IP. Males must be surgically sterile (> 90 days since vasectomy with no viable sperm), or if engaged in sexual relations with a WOCBP, either his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method must be used from Screening until study completion, including the Follow-up period, and 90 days. Males with same-sex partners (abstinence from penile-vaginal intercourse) or are abstinent from heterosexual intercourse are not required to use contraception. Males must not donate sperm from the first dose of IP until at least 90 days after the last dose of IP.

8.Willing and able to comply with all study-related procedures and assessments, including confinement and attending necessary visits to the CRU.

Exclusion Criteria:

1. Has history of febrile illness or evidence of active infection within 14 days prior to the first dose of IP.
2. Substance abuse-related disorder or a history of drug, and/or substance abuse deemed significant by the Investigator. Positive drug screen at Screening, Day 1 for Part D/Part D2 (Period1) and Day -1 for other parts. The test could be repeated once at the discretion of Investigator/designee.
3. Has consumed more than 14 units of alcohol per week in the 3 months prior to signing the ICF (1 unit = 360 mL of beer with an alcohol content of 5%, or 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine with an alcohol content of 12%), or has a positive alcohol breath test (breath alcohol concentration > 0.0 mg/100 mL) at Screening, Day 1 for Part D/Part D2 (Period1) and Day -1 for other parts, or unable to abstain from alcohol during the trial period. The test could be repeated once at the discretion of the Investigator/designee.
4. History of alcohol allergy.
5. Has excessively used nicotine products (average daily smoking of more than 5 cigarettes) within the 3 months prior to Screening or refuse to abstain from smoking during the trial or has a positive nicotine/cotinine test at Day 1 for Part D/Part D2 (Period 1) and Day -1 for other parts.
6. Participated in any other investigational trials or has been exposed to other investigational drugs within 28 days or 5 half-lives of the previously administered investigational drug (date derived from last study procedure [blood collection or dosing] of previous trial), whichever is longer, prior to admission to the CRU.
7. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody at Screening.
8. Donation of blood or significant blood loss ≥ 400 mL in 1 month prior to the first IP administration, has received a blood transfusion or used blood products within 1 month prior to first dosing, or plan to donate blood during this trial or within 1 month after the last IP administration.
9. Plasma donation within 14 days prior to the first administration of IP.
10. Has used any medication within 14 days prior to the first IP administration that the Investigator considers may affect the PK evaluation of the study drug (including prescription drugs, over-the-counter drugs, herbal medicines, functional vitamins, dietary supplements, etc.).
11. History of previous QTc prolongation, or clinically significant abnormal ECG finding at Screening:

    1. Heart rate 45 to 100 beats per minute.
    2. PR 120 to 220 msec.
    3. QRS < 120 msec.
    4. Subjects with parameters outside the ranges of exclusion criteria 12a to 12c should be excluded from the study.
    5. QTcF ≥ 450 msec for males or QTcF ≥ 470 msec for females (confirmed by repeated examinations).
    6. Long QT syndrome.
    7. Use of concomitant medications that are known to prolong QT/QTc.
    8. Abnormal ECG findings as judged by the Investigator.
12. Has liver disease or clinically significant liver impairment at Screening (e.g., aspartate aminotransferase [AST], alanine aminotransferase [ALT], or total bilirubin > 1.5 times the upper limit of normal [ULN]).
13. Has had major surgery within 6 months prior to the Screening, or plan to have any surgeries during their participation in trial.
14. Has any disease or condition that may interfere with the absorption/distribution/metabolism/excretion of the study drug, in the opinion of the Investigator (e.g., dysphagia, gastrointestinal diseases, cholecystectomy).
15. Presence of diseases such as migraine, cardiovascular, liver, endocrine, gastrointestinal, metabolic, neurological, pulmonary, endocrine, psychiatric, or oncological history, or any other evidence deemed to be clinically significant by the Investigator and that may pose a risk to the safety of the subject or interfere with the conduct, progress, or completion of the study.
16. Previous or suspected history of hypersensitivity or allergic reactions to the active ingredients of the study drug or other drugs and food.
17. Consumption of foods or juices containing cranberries or pineapples, Seville oranges, grapefruit, pomegranate or caffeine (xanthine-containing products) for 48 hours prior to each dose and remain restricted until the end of PK collection on each dosing day for Part D and before the start of dosing until after collection of the final PK for other Parts, unless deemed acceptable by the Investigator.
18. Subjects with other factors deemed ineligible to participate in the trial by the Investigator.
19. Subjects who are excessively sensitive to cold pain (PTT < 10 seconds) or who tolerate it too long (PTT > 96 seconds) will be excluded from
20. Part D.Part D/Part D2 ONLY; Subjects who are excessively sensitive to cold pain (defined as a PTT < 10 seconds) or who tolerate cold pain (defined as a PTT > 96 seconds) will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of FZ008-145 solution by number of adverse events (AEs) and treatment-emergent adverse events (TEAEs) | up to 14 days post first dose administration
  Safety of FZ008-145 solution is assessed by the incidence, nature, and severity of adverse events (AEs) and treatment-emergent adverse events (TEAEs) following administration of FZ008-145 solution. AEs and TEAEs are collected from the time of dosing through the end of the study and are summarized by number of participants experiencing at least one event.
To assess the safety of FZ008-145 tablet by number of adverse events (AEs) and treatment-emergent adverse events (TEAEs) | up to 14 days post first dose administration
  Safety of FZ008-145 solution is assessed by the incidence, nature, and severity of adverse events (AEs) and treatment-emergent adverse events (TEAEs) following administration of FZ008-145 solution. AEs and TEAEs are collected from the time of dosing through the end of the study and are summarized by number of participants experiencing at least one event.
Number of participants with changes in laboratory parameters determined as adverse events following oral dose of FZ008-145 solution and FZ008-145 tablet | up to 14 days post first dose administration
  The number of participants experiencing laboratory parameter abnormalities that are assessed as clinically significant and reported as adverse events (AEs) or treatment-emergent adverse events (TEAEs) following oral administration of FZ008-145 solution or FZ008-145 tablet.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  Cmax- Maximum plasma concentration
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  Tmax- Time taken for maximum concentration
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  AUC0-last- Area under curve from 0 to last
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  AUC0-inf- Area under curve from 0 to infinity
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  t1/2- terminal half-life
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  CL/F- Apparent total body clearance
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 5 days post first dose administration
  Vz/F- Apparent total volume of distribution
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 4 days post first dose administration
  Ae- Amount of analyte that is eliminated in urine
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 4 days post first dose administration
  Fe- Fraction of analyte eliminated in Urine
To evaluate the pharmacokinetics (PK) of FZ008-145 solution and FZ008-145 tablet | Up to 4 days post first dose administration
  CLr- Clearance rate

CONTACTS AND LOCATIONS:
Overall Officials: Shiqun Zhang, Study Director — Guangzhou Fermion Technology Co., LTD
Locations (1):
- CMAX Clinical Research Pty, Adelaide, South Australia, Australia